CLINICAL TRIAL: NCT02515981
Title: New Hampshire Medicaid Wellness Incentive Program
Acronym: NHWIP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Dartmouth-Hitchcock Medical Center (Other)
Collaborators: State of New Hampshire Bureau of Behavioral Health (Unknown)
Responsible Party: Principal Investigator, Sarah Pratt, Medicaid Policy Analyst, Dartmouth-Hitchcock Medical Center
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Health Services Research
Other Study IDs: 23336
Record Dates: First submitted 2015-01-30; First posted 2015-08-05 (Estimated); Last update posted 2019-02-19 (Actual); Status verified 2019-02

CONDITIONS: Tobacco Dependence; Obesity; Mental Illness
Keywords: tobacco dependence; smoking cessation; mental health; cardiovascular disease; obesity
MeSH Terms: conditions — Tobacco Use Disorder; Obesity; Mental Disorders; Smoking Cessation; Psychological Well-Being; Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Incentives (Experimental): Participants randomly assigned to the incentive arm, will receive cash incentives for engaging in healthy lifestyle behaviors.
  Interventions: Behavioral: NH Medicaid Incentives Program
- No Incentives (Experimental): Participants randomly assigned to the no incentives arm, will not receive cash incentives for engaging in healthy lifestyle behaviors.
  Interventions: Behavioral: NH Medicaid Incentives Program

INTERVENTIONS:
Behavioral: NH Medicaid Incentives Program

SUMMARY:
The New Hampshire Medicaid Wellness Incentive Program (WIP) will address both the health disparity and increased costs by providing incentivized health promotion programs to overweight or obese and/or tobacco-smoking Medicaid beneficiaries receiving services at New Hampshire's 10 regional Community Mental Health Centers (CMHCs).

DETAILED DESCRIPTION:
In the New Hampshire Medicaid Wellness Incentive Program, multiple program options will fall into two categories: (1) Supported Fitness and Weight Management and (2) Supported Smoking Cessation. Eligible participants are able to participate in 1 or both of the programs. The program options for Supported Fitness and Weight Management are: 1. Fitness Club Membership for 12 months, 2. Fitness Club Membership plus weekly meetings with a Health Mentor for 12 months (In SHAPE), 3. Weight Watchers Membership for 12 months, 4. In SHAPE plus Weight Watchers for 12 months. The options for Supported Smoking Cessation are: 1. Prescriber meeting to discuss smoking cessation treatment options, 2. Prescriber meeting plus NH State Tobacco Helpline, 3. Prescriber meeting plus Telephone-based Cognitive Behavioral Therapy for Smoking Cessation. Vouchers for memberships to community fitness centers and formal weight loss programs will be provided, as well as incentives for participation and positive outcomes. An equipoise stratified randomization design will be used to preserve the research benefits of randomization while maintaining the highly valued opportunity for consumer choice. Research assessments will be conducted at baseline, 3 months, 6 months, 9 months, and 12 months.

ELIGIBILITY:
Inclusion Criteria for smoking intervention and weight management intervention:

* Participants must be Medicaid recipients receiving mental health treatment at one of the participating study sites in New Hampshire.
* 18 years or older

Additional Inclusion Criteria for smoking intervention only:

*Smoking 5 or more cigarettes a day or a carbon monoxide level of 5 or higher at screening.

Additional Inclusion Criteria for weight management only:

*Body Mass Index of 30 or higher or 25 or higher and sedentary lifestyle.

Exclusion Criteria for both interventions:

* Diagnosis of dementia or terminal illness (expected to result in death in 1 year or less)
* Nursing home
* Inability to speak or understand English

Additional exclusion Criteria for weight management only:

* Previous participation in the In SHAPE program
* Active eating disorder diagnosis
* Pregnancy

Additional exclusion Criteria for smoking intervention only:

*Active alcohol or drug dependence with use in the past 30 days

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2800 (Estimated)
Dates: Start 2012-05; Primary Completion 2016-04 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Change in Weight | Baseline, 3 months, 6 months, 9 months, 12 months and 1 year post program follow up
  Weight obtained using a scale at each assessment.
Change in the 6 minute walk test | Baseline, 3 months, 6 monhts, 9 months, 12 months, and 1 year post program completion follow up
  Each participant walks as many ft as possible at a brisk pace. The amount of feet covered in 6 minutes is documented.
Change in Days of Abstinence-Timeline follow back interview for tobacco smokers | Baseline, 3 months, 6 months, 9 months, 12 months, and 1 year post program completion follow up
  A timeline follow back interview is completed for the smoking cessation intervention to identify days of abstinence within the assessment period as well as amount of cigarettes smoked.
Change in Carbon Monoxide Level | Baseline, 3 months, 6 months, 9 months, 12 months, and 1 year post program completion follow up
  At each assessment and during the incentive quit cycles, carbon monoxide level is measured to confirm smoking abstinence or not.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah I Pratt, PhD, Study Director — Dartmouth-Hitchcock Medical Center; Kelley Capuchino, Principal Investigator — State of New Hampshire, Department of Health and Human Services
Locations (12):
- United States (12):
  - New Hampshire Hospital, Concord, New Hampshire
  - Riverbend Community Mental Health Center, Concord, New Hampshire
  - Center for Life Management, Derry, New Hampshire
  - Community Partners, Dover, New Hampshire
  - Mondadnock Family Services, Keene, New Hampshire
  - West Central Behavioral Health Care, Lebanon and Claremont, New Hampshire
  - Northern Human Services, Littleton and Conway, New Hampshire
  - The Mental Health Center of Greater Manchester, Manchester, New Hampshire
  - Greater Nashua Mental Health Center at Community Council, Nashua, New Hampshire
  - Harbor Homes, Nashua, New Hampshire
  - Genesis Behavioral Heatlh, Plymouth and Laconia, New Hampshire
  - Seacoast Mental Health Center, Portsmouth, New Hampshire

REFERENCES:
- [Derived] Pratt SI, Ferron JC, Wolfe R, Xie H, Brunette M, Santos M, Williams G, Bartels S, Jue K, Capuchino K. Healthy choices, healthy changes: A randomized trial of incentives to promote healthy eating and exercise in people with schizophrenia and other serious mental illnesses. Schizophr Res. 2023 May;255:1-8. doi: 10.1016/j.schres.2023.03.007. Epub 2023 Mar 16. PMID 36933290
- [Derived] Bianco CL, Pratt SI, Ferron JC, Brunette MF. Electronic Cigarette Use During a Randomized Trial of Interventions for Smoking Cessation Among Medicaid Beneficiaries with Mental Illness. J Dual Diagn. 2019 Jul-Sep;15(3):184-191. doi: 10.1080/15504263.2019.1620400. Epub 2019 Jun 6. PMID 31169077
- [Derived] Brunette MF, Pratt SI, Bartels SJ, Scherer EA, Sigmon SC, Ferron JC, Santos M, Williams GE, Kosydar S, Wolfe RS, Lotz D, Capuchino K. Randomized Trial of Interventions for Smoking Cessation Among Medicaid Beneficiaries With Mental Illness. Psychiatr Serv. 2018 Mar 1;69(3):274-280. doi: 10.1176/appi.ps.201700245. Epub 2017 Nov 15. PMID 29137560